CLINICAL TRIAL: NCT06610474
Title: Evaluation of an Online Prostate Cancer Screening Decision Aid
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: David Siegel (U.S. Federal Agency)
Collaborators: ICF Macro, Inc. (Other)
Responsible Party: Sponsor-Investigator, David Siegel, Medical Officer, Division of Cancer Prevention and Control, Principal Investigator, Centers for Disease Control and Prevention
Organization: Centers for Disease Control and Prevention (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 2023-030
Record Dates: First submitted 2024-09-20; First posted 2024-09-24 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Prostate Cancer
Keywords: Decision Aid
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Talk to Nathan (Experimental): Participants in this arm will use the online "Talk to Nathan about Prostate Cancer Screening" decision aid before their clinic visit.
  Interventions: Behavioral: Use of the online "Talk to Nathan about Prostate Cancer" decision aid
- Standard decision aid (Active Comparator): Participants in this arm will use a standard decision aid before their clinic visit.
  Interventions: Behavioral: Use of a standard prostate cancer screening decision aid
- Standard education materials (Active Comparator): Participants in this arm will use standard education materials before their clinic visit.
  Interventions: Behavioral: Use of standard prostate cancer education materials

INTERVENTIONS:
Behavioral: Use of the online "Talk to Nathan about Prostate Cancer" decision aid — This decision aid is publicly available at this website in both English or Spanish: https://www.cdc.gov/prostate-cancer/talk-to-nathan/index.html
  Arms: Talk to Nathan
Behavioral: Use of a standard prostate cancer screening decision aid — The standard decision aid is available here and will be used in either English or Spanish: https://massclearinghouse.ehs.state.ma.us/PROG-CANC/CA1382kit.html
  Arms: Standard decision aid
Behavioral: Use of standard prostate cancer education materials — The standard education materials are available from the National Cancer Institute (NCI) website in English or Spanish: https://www.cancer.gov/types/prostate/patient/prostate-screening-pdq
  Arms: Standard education materials

SUMMARY:
The goal of this clinical trial is to learn if the online, simulated human "Talk to Nathan About Prostate Cancer Screening" decision aid (https://www.cdc.gov/prostate-cancer/talk-to-nathan/index.html) is effective in helping patients decide about prostate cancer screening. The main questions it aims to answer are:

* Is using the "Talk to Nathan About Prostate Cancer Screening" decision aid effective in improving knowledge, overcoming health literacy barriers, and resolving decisional conflict compared to a standard decision aid or standard education materials?
* What are the barriers and best practices for incorporating Talk to Nathan About Prostate Cancer Screening into the flow of primary care practice?

Researchers will compare "Talk to Nathan About Prostate Cancer Screening" to a standard decision aid and to standard prostate cancer screening education materials to test the effectiveness of using "Talk to Nathan About Prostate Cancer Screening."

Participants will:

* Use "Talk to Nathan About Prostate Cancer Screening," use a standard decision aid, or use standard education materials about prostate cancer screening
* Visit the primary care clinic for follow-up
* Complete surveys as part of the clinical trial

DETAILED DESCRIPTION:
Goal of the project: To conduct a randomized controlled trial (RCT) to determine if CDC's online, simulated, human decision aid module, Talk to Nathan About Prostate Cancer Screening (treatment arm), is effective in improving knowledge, overcoming health literacy barriers, and resolving decisional conflict compared to a standard decision aid (control arm 1) and standard education materials (control arm 2). Also, to identify barriers and best practices for incorporating Talk to Nathan About Prostate Cancer Screening into the flow of primary care practice.

Intended use of the resulting data: To measure evaluation outcomes, understand how to help men make decisions about the harms and benefits of prostate cancer screening that are in line with the patient's individual values and preferences, and make recommendations for improving the Talk to Nathan About Prostate Cancer Screening decision aid and incorporating it into primary care practice.

Methods to be used to collect: The RCT is a three-group parallel design with one treatment arm and two control arms. Data will be collected from all arms using a pre-exposure survey, a post-exposure survey, and a post-clinic visit survey. The treatment arm will also complete a usability survey and a subset of the treatment arm will be invited to participate in user experience interviews. Health care providers at the four participating clinics will complete a short survey prior to executing the three-arm study and interviews will be conducted at the close of the study with study coordinators from the four participating clinics.

The subpopulation to be studied: For the pre- and post-surveys, the usability survey, and the user experience interviews, the subpopulation is men aged 55-69 years. For the provider survey, the subpopulation is primary care providers who practice within the four clinics participating in the study. For the clinic coordinator interviews, the subpopulation is the study coordinators from the four participating clinics.

How data will be analyzed: For quantitative survey data: intention-to-treat analysis; repeated measures analysis of variance across assessment time points; ordinary least squares regression; complier-average causal effect (CACE) approach to calculate treatment effect; maximum likelihood and Bayesian inferential methods for CACE. For qualitative data from the surveys and interviews: We will identify and analyze themes, patterns, and inter-relationships relevant to the evaluation questions for this study.

ELIGIBILITY:
Inclusion Criteria:

* Male.
* Aged 55-69 years.
* Scheduled for an upcoming health exam.
* Has access to the internet.
* Has a valid email address or valid mobile phone number with SMS capabilities.
* Speaks and reads English or Spanish.

Exclusion Criteria:

* Refuses to participate.
* Currently has urinary tract symptoms (i.e., difficulty starting urination; weak or interrupted flow of urine; urinating often, especially at night; trouble emptying the bladder completely; pain or burning during urination; blood in the urine or semen; pain in the back, hips, or pelvis that doesn't go away; or painful ejaculation).
* Prior history of prostate cancer.
* Scheduled for, undergoing, or has had a prostate biopsy.
* A previous PSA score is contained in the patient's health record and it is greater than or equal to 4 ng/mL and/or a very suspicious digital rectal exam (DRE) result (defined as the presence of significant induration, nodularity, or asymmetry).
* Patient has a terminal illness, significant psychiatric comorbidity (identified by clinic coordinator), cognitive deficits, or reports of ongoing substance misuse.

Ages: 55 Years to 69 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 510 (Estimated)
Dates: Start 2024-11-27 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Measure of changes in decisional conflict | Immediately after clinical encounter with provider
  Assessment by participant survey

SECONDARY OUTCOMES:
Measure of prostate cancer knowledge | Immediately after clinical encounter with provider
  Assessment by participant survey
Measure of autonomous decision-making | Immediately after clinical encounter with provider
  Assessment by participant survey

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - East Northport Medical Care, East Northport, New York
  - Camino, Charlotte, North Carolina
  - Alliance Medical Ministry, Raleigh, North Carolina
  - Clemson Rural Health, Clemson, South Carolina

IPD SHARING:
Plan to Share IPD: Yes
In development.